CLINICAL TRIAL: NCT04020211
Title: HF10 Therapy for the Treatment of Chronic, Focal, Neuropathic Pain Following Orthopedic Surgical Intervention of the Knee(s) - A Multicenter, Prospective Clinical Trial
Brief Title: HF10 Treatment of Chronic Knee Pain
Acronym: CPSP-3
Status: Terminated | Type: Observational
Why Stopped: Limited Enrollment
Sponsor: Nevro Corp (Industry)
Responsible Party: Sponsor
Other Study IDs: CA2018-5 US CPSP-3
Record Dates: First submitted 2019-04-09; First posted 2019-07-15 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain Post-Procedural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- HF10: SCS stimulation with HF10 therapy
  Interventions: Device: Senza HF10 Therapy

INTERVENTIONS:
Device: Senza HF10 Therapy — Senza 10kHz Spinal Cord Stimulation
  Other Names: Nevro Senza Spinal Cord Stimulation (SCS)

SUMMARY:
This is a multi-center study where patients who meet the eligibility criteria will be treated with HF10 therapy for their chronic knee pain post-orthopedic surgery. The primary endpoint will be assessed at 3 months, but observational assessments will continue until study completion at 12 months following implant.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have been diagnosed with chronic, focal, neuropathic pain following orthopedic surgery(ies) of the knee(s).
2. Average pain intensity (over a period of 7 days) of ≥5 out 10 cm on the Visual Analog Scale (VAS) in the primary area of pain at enrollment.
3. Have a score of at least 4 out of 10 in Douleur Neuropathique 4 (DN4) questionnaire at the time of enrollment or eligibility verification.
4. Deemed not to have surgical loosening or other complications from the surgery that affect the stability of the knee.
5. Have stable neurological status measured by motor, sensory and reflex function as determined by the investigator.
6. Be on stable pain medications, as determined by the Investigator, for at least 28 days prior to assessing pain intensity as described in inclusion criterion #2, and be willing to stay on those medications with no dose adjustments until activation of the permanently implanted SCS device.

Key Exclusion Criteria:

1. Have radiculopathy or radicular leg pain resulting from failed back surgery.
2. Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator (such as primary headache diagnosis or fibromyalgia).
3. Have a current diagnosis of a progressive neurological disease such as multiple sclerosis (MS), chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, brain or spinal cord tumor, central deafferentation syndrome, acute herniating disc, severe spinal stenosis and brachial plexus avulsion as determined by the Investigator.
4. Have a current diagnosis or condition such as a coagulation disorder, bleeding diathesis, platelet dysfunction, progressive peripheral vascular disease or uncontrolled diabetes mellitus that presents excess risk for performing the procedure as determined clinically by the Investigator.
5. Have any prior experience with SCS.
6. Have objective evidence of epidural scarring and/or any signs or symptoms of myelopathy as determined by the investigator.
7. Be benefitting from an interventional procedure to treat their trunk or limb pain (Subjects should be enrolled at least 30 days from last benefit).
8. Have an existing drug pump and/or another active implantable device such as a pacemaker.
9. Be involved in an injury claim under current litigation.
10. Have an active or unsettled worker's compensation claim.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the eligibility criteria will be treated with HF10 therapy for their chronic knee pain post-orthopedic surgery.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Responders and Improvement in Oxford Knee Score (OKS) | 3 months
  The OKS is a patient self-completion patient reported outcome containing 12 questions on activities of daily living with a recall period of 4 weeks. The OKS has been developed and validated specifically to assess function and pain after total knee replacement. The higher the score indicates improvement. The proportion of implanted subjects who are responders (achieved ≥ 50% pain relief) to HF10 therapy for treatment of their chronic, post-surgical knee pain or reporting at least a 4-point improvement in their Oxford Knee Score (OKS).

SECONDARY OUTCOMES:
Change in Disability and Functioning | 3, 6, and 12 months
  Percentage and average change from Baseline in Oxford Knee Score
Change in Functioning | 3 and 12 months
  Average change in walking distance assessed by 6-minute Walk Test
Change in Functioning | 3 and 12 months
  Change in Global Assessment of Functioning
Change in pain relief as measured by the Visual Analog Scale (VAS) | 3 and 12 months
  Percentage and average change from Baseline in knee pain intensity
Change from baseline in pain experience: Short-Form McGill Pain Questionnaire (SF-MPQ-2) scores | 3 and 12 months
  The Short Form McGill Pain Questionnaire version 2 (SF-MPQ-2, hereafter referred to as MPQ) is a well validated and widely used questionnaire used to measure the major symptoms of pain. Subjects will be asked to rate the intensity of each of 22 pain descriptors from 0 (do not experience, or none) to 10 (worst possible) at follow-up visits outlined in the schedule of events.
  Four subscale scores (continuous pain, intermittent pain, predominantly neuropathic pain, and affective descriptors) and a total score will be calculated. The lower the score indicates improvement (less interference from pain). Each subject's baseline scores will be compared to the scores at study visits. Mean change from baseline will be calculated for the entire cohort.
  Percentage and average change from Baseline in Short-Form McGill Pain Questionnaire (SF-MPQ-2) scores
Global Impression of Change | 3 and 12 months
  Subject's impression of change in overall health condition as measured by the Patient and Clinician Global Impression of Change
Change in Quality of Life as measured by the EuroQol five-dimensional questionnaire (EQ-5D-5L) | 3 and 12 months
  The 5-level EQ-5D version (EQ-5D-5L) uses a 2-part assessment: a descriptive one and a visual analog scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The higher the score indicates an improved in quality of life. Change from Baseline in health-related quality of life evaluation
Change in Sleep as measured by the Pain and sleep Questionnaire (PSQ) | 3 and 12 months
  PSQ is an eight-item questionnaire developed to assess the impact of pain on sleep. PSQ-3 is a subset of PSQ, consisting of questions 1, 4 and 5 and has been validated to assess impact of chronic pain on sleep. The lower the score indicates improvement by less interference of sleep from pain. Change from baseline in 3-item pain and sleep questionnaire
Medication | 3 and 12 months
  Change from baseline in opioid equivalent medication usage
Safety profile: Incidence of AEs over time | 3, 6 and 12 months
  Incidence of AEs over time
Safety profile: Neurological assessment over time by a physician and exam | 3, 6 and 12 months
  Neurologic status includes testing for gross motor, sensory and appropriate reflex functions, which will be characterized as improved, maintained, or a deficit as compared with baseline status as follows: A clinically meaningful neurological improvement is defined as a significant persistent improvement in neurological function that impacts subject's well-being is attributable to a neurological finding; and is new or improved as compared with the baseline assessment. A clinically meaningful neurological deficit is defined as a stimulation-related significant persistent abnormality in neurological function that impacts subject's well-being is attributable to a neurological finding; and is new or worsened as compared with the baseline assessment. If neither a clinically meaningful neurological improvement nor a clinically meaningful neurological deficit is observed, then neurologic status is maintained.

CONTACTS AND LOCATIONS:
Overall Officials: David Caraway, MD, Study Director — Chief Medical Officer
Locations (1):
- Pain Management, Greenfield, Wisconsin, United States